CLINICAL TRIAL: NCT02360605
Title: Health Literacy Interventions to Overcome Disparities in CRC Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Northwestern University (Other); Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RSG-13-021-01 - CPPB; RSG-13-021-01 - CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; low literacy; community clinics; Fecal Immunochemical Test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- automated telephone reminder arm (Active Comparator): Patients will receive Health literacy appropriate education and demonstration of FIT kits with simplified instructions. Patients will receive reminders to complete their FIT screening kits by an automated call.
  Interventions: Behavioral: automated telephone reminder; Behavioral: Health literacy appropriate education and demonstration
- prevention coordinator arm (Active Comparator): Patients will receive Health literacy appropriate education and demonstration of FIT kits with simplified instructions.Patients will receive reminders to complete their FIT screening kits by a prevention coordinator.
  Interventions: Behavioral: prevention coordinator; Behavioral: Health literacy appropriate education and demonstration

INTERVENTIONS:
Behavioral: automated telephone reminder — The patients will be contacted at 4 weeks and again at 8 weeks if they have not returned the FIT. ATR will remind the patient of the importance of completing and returning the FIT results and encourage screening completion. There will also be an option where the patient can request another FIT kit be mailed to them, one to hear information on common problems with FIT completion or how to call the clinic if they have questions. Years 2 and 3: 12 months after patients returned their initial FIT (or if they did not return the FIT, 12 months after enrollment) they will be mailed a friendly letter to remind them that it is time for their annual CRC screening and that a FIT kit will be mailed the following week. During the following week the patients will be mailed the FIT kit with addressed stamped envelope and the educational pamphlet they received at enrollment. For follow-up ATR calls, we will use the same protocol as described for the initial screening. Same procedure for year 3.
  Arms: automated telephone reminder arm
Behavioral: prevention coordinator — The patients will be contacted at 4 weeks and again at 8 weeks if they have not returned the FIT by a prevention coordinator (PC). PC will call to encourage completion and ascertain any barriers to completion. The PCs will use Health Literacy and motivational interviewing techniques described in the training section to enhance understanding and confidence and reduce ambivalence to completing and returning the FIT. Years 2 and 3: 12 months after patients returned their initial FIT (or if they did not return the FIT, 12 months after enrollment) they will be mailed a friendly letter to remind them that it is time for their annual CRC screening and that a FIT kit will be mailed the following week. During the following week the patients will be mailed the FIT kit with addressed stamped envelope and the educational pamphlet they received at enrollment. For follow-up PC calls, we will use the same protocol as described for the initial screening. Same procedure for year 3.
  Arms: prevention coordinator arm
Behavioral: Health literacy appropriate education and demonstration — The Research Assistant (RA) will employ health literacy communication principles in providing a CRC recommendation and brief screening information using the CRC pamphlet and a FIT kit with simplified instructions and accompanying self-addressed, stamped envelope. A scripted message and illustrations will model what the patient needs to do to complete the FIT. The RA will appropriately demonstrate, using the kit, and will suggest patients show the pamphlet and FIT kit to their provider that day and talk to them about screening. Annual screening will be further emphasized at enrollment by giving patients an empowering message about the benefits of completing a FIT annually and telling them they will be mailed a reminder letter and FIT kit and receive outreach phone calls in 12 and 24 months for the next two years as well as a post survey and satisfaction interview over the phone at 6 months.

SUMMARY:
In the proposed project the investigators will evaluate two different follow-up approaches to improve low income patients' completion of initial and annual colorectal cancer (CRC) screening using the Fecal Immunochemical Test (FIT), the most sensitive FOBT. The purpose of this study is to compare the effectiveness of two distinct follow-up strategies to promote CRC screening: a prevention coordinator (PC) approach vs. an automated telephone reminder (ATR) system. The investigators will adapt a successful intervention tested in the Health Literacy and Cancer Screening Project by adding a follow-up strategy to the health literacy intervention. Specific Aims: The investigators Primary Aims are to: 1. Compare the effectiveness of the PC and ATR strategies to improve initial and repeat CRC screening. 2. Compare the cost effectiveness of the PC and ATR strategies for initial and repeat CRC screening. The investigators Secondary Aims are to: 3. Conduct a process evaluation of both follow-up strategies to investigate implementation and barriers 4. Determine if the effects of either strategy vary by patients' literacy skills. 5. Explore patient characteristics associated with CRC screening knowledge, beliefs, self-efficacy, and compliance over time between study arms.

DETAILED DESCRIPTION:
The investigators objective is to compare the effectiveness of two distinct follow-up strategies to promote colorectal cancer screening: a prevention coordinator (PC) approach vs. an automated telephone reminder (ATR) system. The investigators will adapt a successful intervention tested in the Health Literacy and Cancer Screening Project [R01CA115869] by adding a follow-up strategy to the health literacy intervention. In the proposed project the investigators will evaluate two different follow-up approaches to improve low income patients' completion of initial and annual CRC screening using Fecal Immunochemical Test (FIT).

Substantial evidence shows that routine screening can prevent colorectal cancer (CRC) or detect it at an early stage, reducing related mortality. While overall CRC screening rates in the US are increasing, rates remain persistently low among uninsured and low-income individuals, those with fewer years of education, and racial/ethnic minorities. Low health literacy has been linked to cancer screening noncompliance, higher rates of advanced stage of presentation of disease and health disparities. In response, the Department of Health and Human Services has called for health information and services that are accurate, accessible, and actionable as well as culturally appropriate.

This study will implement a two-arm, randomized controlled trial with low income, underinsured patients in federally qualified health centers (FQHCs) to evaluate and compare the effectiveness of PC and ATR follow-up strategies to increase CRC screening. All patients recruited to the study will receive evidence-based, literacy appropriate screening materials developed using health literacy 'best practices' and a simplified FIT kit. Use of these materials has been shown to significantly increase CRC screening rates in the investigators ongoing study. Patients will be randomized to receive either: 1) the PC follow-up strategy, in which a PC personally reminds patients to complete and mail FIT kits, and perceived barriers to screening are discussed and addressed; or 2) the ATR follow-up strategy, in which an automated system electronically encourages patients to complete and mail FIT kits using plain language messages. The effectiveness of these two approaches will be compared at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. a patient of the identified clinics,
2. age 50 to 75 (based on American Cancer Society (ACS) guidelines), and
3. can speak and understand English

Exclusion Criteria:

1. previous history of cancer other than non-melanoma skin cancer,
2. up-to-date with CRC screening according to ACS guidelines (FOBT every year, sigmoidoscopy every 5 years, or colonoscopy every 10 years),
3. a first relative family history that requires a more complete history and possible colonoscopy because of their risk factor (these patients will be referred to their provider for follow-up),
4. an uncorrectable hearing or visual impairment, or
5. too ill to participate.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2015-02; Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Health Sciences Center, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levin B, Lieberman DA, McFarland B, Andrews KS, Brooks D, Bond J, Dash C, Giardiello FM, Glick S, Johnson D, Johnson CD, Levin TR, Pickhardt PJ, Rex DK, Smith RA, Thorson A, Winawer SJ; American Cancer Society Colorectal Cancer Advisory Group; US Multi-Society Task Force; American College of Radiology Colon Cancer Committee. Screening and surveillance for the early detection of colorectal cancer and adenomatous polyps, 2008: a joint guideline from the American Cancer Society, the US Multi-Society Task Force on Colorectal Cancer, and the American College of Radiology. Gastroenterology. 2008 May;134(5):1570-95. doi: 10.1053/j.gastro.2008.02.002. Epub 2008 Feb 8. PMID 18384785
- [Background] Edwards BK, Ward E, Kohler BA, Eheman C, Zauber AG, Anderson RN, Jemal A, Schymura MJ, Lansdorp-Vogelaar I, Seeff LC, van Ballegooijen M, Goede SL, Ries LA. Annual report to the nation on the status of cancer, 1975-2006, featuring colorectal cancer trends and impact of interventions (risk factors, screening, and treatment) to reduce future rates. Cancer. 2010 Feb 1;116(3):544-73. doi: 10.1002/cncr.24760. PMID 19998273
- [Background] Steinwachs D, Allen JD, Barlow WE, Duncan RP, Egede LE, Friedman LS, Keating NL, Kim P, Lave JR, Laveist TA, Ness RB, Optican RJ, Virnig BA. National Institutes of Health state-of-the-science conference statement: Enhancing use and quality of colorectal cancer screening. Ann Intern Med. 2010 May 18;152(10):663-7. doi: 10.7326/0003-4819-152-10-201005180-00237. Epub 2010 Apr 13. No abstract available. PMID 20388702
- [Background] Taplin SH, Haggstrom D, Jacobs T, Determan A, Granger J, Montalvo W, Snyder WM, Lockhart S, Calvo A. Implementing colorectal cancer screening in community health centers: addressing cancer health disparities through a regional cancer collaborative. Med Care. 2008 Sep;46(9 Suppl 1):S74-83. doi: 10.1097/MLR.0b013e31817fdf68. PMID 18725837
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: colorectal cancer screening among adults aged 50-75 years - United States, 2008. MMWR Morb Mortal Wkly Rep. 2010 Jul 9;59(26):808-12. PMID 20613704
- [Background] Davis TC, Dolan NC, Ferreira MR, Tomori C, Green KW, Sipler AM, Bennett CL. The role of inadequate health literacy skills in colorectal cancer screening. Cancer Invest. 2001;19(2):193-200. doi: 10.1081/cnv-100000154. PMID 11296623
- [Background] Davis TC, Williams MV, Marin E, Parker RM, Glass J. Health literacy and cancer communication. CA Cancer J Clin. 2002 May-Jun;52(3):134-49. doi: 10.3322/canjclin.52.3.134. PMID 12018928
- [Background] Dolan NC, Ferreira MR, Davis TC, Fitzgibbon ML, Rademaker A, Liu D, Schmitt BP, Gorby N, Wolf M, Bennett CL. Colorectal cancer screening knowledge, attitudes, and beliefs among veterans: does literacy make a difference? J Clin Oncol. 2004 Jul 1;22(13):2617-22. doi: 10.1200/JCO.2004.10.149. PMID 15226329
- [Background] Burt RW. Strategies for colon cancer screening with considerations of cost and access to care. J Natl Compr Canc Netw. 2010 Jan;8(1):2-5. doi: 10.6004/jnccn.2010.0002. No abstract available. PMID 20064288
- [Background] O'Malley AS, Beaton E, Yabroff KR, Abramson R, Mandelblatt J. Patient and provider barriers to colorectal cancer screening in the primary care safety-net. Prev Med. 2004 Jul;39(1):56-63. doi: 10.1016/j.ypmed.2004.02.022. PMID 15207986
- [Background] Lasser KE, Ayanian JZ, Fletcher RH, Good MJ. Barriers to colorectal cancer screening in community health centers: a qualitative study. BMC Fam Pract. 2008 Feb 27;9:15. doi: 10.1186/1471-2296-9-15. PMID 18304342
- [Background] Greiner KA, Born W, Nollen N, Ahluwalia JS. Knowledge and perceptions of colorectal cancer screening among urban African Americans. J Gen Intern Med. 2005 Nov;20(11):977-83. doi: 10.1111/j.1525-1497.2005.00165.x. PMID 16307620
- [Background] Davis TC, Arnold CL, Rademaker AW, Platt DJ, Esparza J, Liu D, Wolf MS. FOBT completion in FQHCs: impact of physician recommendation, FOBT information, or receipt of the FOBT kit. J Rural Health. 2012 Summer;28(3):306-11. doi: 10.1111/j.1748-0361.2011.00402.x. Epub 2012 Jan 24. PMID 22757955
- [Background] Arnold CL, Rademaker A, Bailey SC, Esparza JM, Reynolds C, Liu D, Platt D, Davis TC. Literacy barriers to colorectal cancer screening in community clinics. J Health Commun. 2012;17 Suppl 3(0 3):252-64. doi: 10.1080/10810730.2012.713441. PMID 23030574
- [Background] Khankari K, Eder M, Osborn CY, Makoul G, Clayman M, Skripkauskas S, Diamond-Shapiro L, Makundan D, Wolf MS. Improving colorectal cancer screening among the medically underserved: a pilot study within a federally qualified health center. J Gen Intern Med. 2007 Oct;22(10):1410-4. doi: 10.1007/s11606-007-0295-0. Epub 2007 Jul 26. PMID 17653808
- [Background] Baron RC, Melillo S, Rimer BK, Coates RJ, Kerner J, Habarta N, Chattopadhyay S, Sabatino SA, Elder R, Leeks KJ; Task Force on Community Preventive Services. Intervention to increase recommendation and delivery of screening for breast, cervical, and colorectal cancers by healthcare providers a systematic review of provider reminders. Am J Prev Med. 2010 Jan;38(1):110-7. doi: 10.1016/j.amepre.2009.09.031. PMID 20117566
- [Background] Zapka J. Innovative provider- and health system-directed approaches to improving colorectal cancer screening delivery. Med Care. 2008 Sep;46(9 Suppl 1):S62-7. doi: 10.1097/MLR.0b013e31817fdf57. No abstract available. PMID 18725835
- [Background] Roetzheim RG, Christman LK, Jacobsen PB, Cantor AB, Schroeder J, Abdulla R, Hunter S, Chirikos TN, Krischer JP. A randomized controlled trial to increase cancer screening among attendees of community health centers. Ann Fam Med. 2004 Jul-Aug;2(4):294-300. doi: 10.1370/afm.101. PMID 15335126
- [Background] Myers RE, Sifri R, Hyslop T, Rosenthal M, Vernon SW, Cocroft J, Wolf T, Andrel J, Wender R. A randomized controlled trial of the impact of targeted and tailored interventions on colorectal cancer screening. Cancer. 2007 Nov 1;110(9):2083-91. doi: 10.1002/cncr.23022. PMID 17893869
- [Background] Stokamer CL, Tenner CT, Chaudhuri J, Vazquez E, Bini EJ. Randomized controlled trial of the impact of intensive patient education on compliance with fecal occult blood testing. J Gen Intern Med. 2005 Mar;20(3):278-82. doi: 10.1111/j.1525-1497.2005.40023.x. PMID 15836533
- [Background] Church TR, Yeazel MW, Jones RM, Kochevar LK, Watt GD, Mongin SJ, Cordes JE, Engelhard D. A randomized trial of direct mailing of fecal occult blood tests to increase colorectal cancer screening. J Natl Cancer Inst. 2004 May 19;96(10):770-80. doi: 10.1093/jnci/djh134. PMID 15150305
- [Background] Pignone M, DeWalt DA, Sheridan S, Berkman N, Lohr KN. Interventions to improve health outcomes for patients with low literacy. A systematic review. J Gen Intern Med. 2005 Feb;20(2):185-92. doi: 10.1111/j.1525-1497.2005.40208.x. PMID 15836553
- [Background] Steele RJ, Kostourou I, McClements P, Watling C, Libby G, Weller D, Brewster DH, Black R, Carey FA, Fraser C. Effect of repeated invitations on uptake of colorectal cancer screening using faecal occult blood testing: analysis of prevalence and incidence screening. BMJ. 2010 Oct 27;341:c5531. doi: 10.1136/bmj.c5531. PMID 20980376
- [Background] DeFrank JT, Rimer BK, Gierisch JM, Bowling JM, Farrell D, Skinner CS. Impact of mailed and automated telephone reminders on receipt of repeat mammograms: a randomized controlled trial. Am J Prev Med. 2009 Jun;36(6):459-67. doi: 10.1016/j.amepre.2009.01.032. Epub 2009 Apr 11. PMID 19362800
- [Background] Lee JK, Reis V, Liu S, Conn L, Groessl EJ, Ganiats TG, Ho SB. Improving fecal occult blood testing compliance using a mailed educational reminder. J Gen Intern Med. 2009 Nov;24(11):1192-7. doi: 10.1007/s11606-009-1087-5. Epub 2009 Sep 23. PMID 19774423
- [Background] Mosen DM, Feldstein AC, Perrin N, Rosales AG, Smith DH, Liles EG, Schneider JL, Lafata JE, Myers RE, Kositch M, Hickey T, Glasgow RE. Automated telephone calls improved completion of fecal occult blood testing. Med Care. 2010 Jul;48(7):604-10. doi: 10.1097/MLR.0b013e3181dbdce7. PMID 20508529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from February 2015-October 2016 in four Federally Qualified Health Centers in rural South Louisiana. Clinic staff asked consecutive patients aged 50 to 75 presenting to the clinic for a scheduled routine primary care visit if they were interested in participating in a CRC screening study.
Groups:
- Automated Telephone Reminder Arm: Patients will receive Health literacy appropriate education and demonstration of FIT kits with simplified instructions. Patients will receive reminders to complete their FIT screening kits by an automated call.
  automated telephone reminder: The patients will be contacted at 4 weeks and again at 8 weeks if they have not returned the FIT. ATR will remind the patient of the importance of completing and returning the FIT results and encourage screening completion. There will also be an option where the patient can request another FIT kit be mailed to them, one to hear information on common problems with FIT completion or how to call the clinic if they have questions.
  Years 2 and 3: 12 months after patients returned their initial FIT (or if they did not return the FIT, 12 months after enrollment) they will be mailed a reminder letter and a FIT kit will be mailed the following week. Follow-up procedure will be the same as year 1.
- Prevention Coordinator Arm: Patients will receive Health literacy appropriate education and demonstration of FIT kits with simplified instructions.Patients will receive reminders to complete their FIT screening kits by a prevention coordinator.
  Prevention coordinator: The patients will be contacted at 4 weeks and again at 8 weeks if they have not returned the FIT by a prevention coordinator (PC). PC will call to encourage completion and ascertain any barriers to completion. The PCs will use Health Literacy and motivational interviewing techniques described in the training section to enhance understanding and confidence and reduce ambivalence to completing and returning the FIT.
  Years 2 and 3: 12 months after patients returned their initial FIT (or if they did not return the FIT, 12 months after enrollment) they will be mailed a friendly reminder letter and then a FIT kit will be mailed the following week. Follow-up calls will follow year 1 procedure.
Period: Overall Study
Arm/Group | Automated Telephone Reminder Arm | Prevention Coordinator Arm
Started | 311 | 309
Completed | 300 | 291
Not Completed | 11 | 18
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Lost to Follow-up | 7 | 8
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: 6 patients withdrew within a day of enrolling and therefore were not included in the CRC analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Automated Telephone Reminder Arm | Prevention Coordinator Arm | Total
Number analyzed (Participants) | 308 | 306 | 614
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (5.9) | 58.6 (6.3) | 58.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 169 | 334
  Male | 143 | 137 | 280
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 210 | 196 | 406
  White | 95 | 109 | 204
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Initial CRC Screening
Description: A patient will be considered screened initially for CRC if he/she completes a FIT within 6 months of study entry.
Time Frame: 6 months after receipt of FIT kit
Measure: Count of Participants; unit: Participants
Groups:
- Prevention Coordinator Arm: Patients will receive Health literacy appropriate education and demonstration of FIT kits with simplified instructions.Patients will receive reminders to complete their FIT screening kits by a prevention coordinator.
  prevention coordinator: patients will be contacted at 4 weeks and again at 8 weeks if they have not returned the FIT by a prevention coordinator (PC). PC will call to encourage completion and ascertain any barriers to completion. The PCs will use Health Literacy and motivational interviewing techniques described in the training section to enhance understanding and confidence and reduce ambivalence to completing and returning the FIT. Years 2 and 3: 12 months after patients returned their initial FIT (or if they did not return the FIT, 12 months after enrollment) they will be mailed a friendly letter to remind them that it is time for their annual CRC screening and that a FIT kit will be mailed the following week. During the following week the patients will be mailed
Arm/Group | Automated Telephone Reminder Arm | Prevention Coordinator Arm
Number analyzed (Participants) | 308 | 306
Participants | 213 | 205
Statistical Analysis 1: Comparison: Automated Telephone Reminder Arm vs Prevention Coordinator Arm; FIT completion rates were defined as the percentage of FIT tests returned. Screening ratios were defined as the PC to AC ratio of FIT completion rates. Multivariate analyses adjusting for age, race, gender, and literacy level were done using generalized linear models. Multivariate analyses adjusting for age, race, gender, and literacy level were done using generalized linear models. A test for interaction between literacy level and study arm were assessed; Test type: Superiority; p = 0.61, Mixed Models Analysis — p-values control for age (in years), race (African American vs Caucasian and Hispanic), gender, and literacy (2 categories) The a priori threshold for statistical significance was p<0.05

2. Primary Outcome: Repeat CRC Screening
Description: Patients in our study will be considered to have completed repeat annual CRC screening if they complete a FIT between 12 and 18 months of previous screen (or baseline interview, if initial FIT was not returned). Year 2 primary outcome is number of participants who return a FIT for 2 years.
Time Frame: between 12 and 18 months of previous screen, 2 years overall
Population: 620 participants enrolled - 6 withdrew the day after enrollment - 614 participants at baseline. Of these, 44 had a positive FIT result and were excluded from the second FIT screening and 2 withdrew after year 1 resulting in a sample size of 568 for the 2nd year screening analysis. All participants who were enrolled were included in the final analysis with the exception of the 44 with a positive FIT test in Year 1 and the 2 lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Automated Telephone Reminder Arm: Years 2 and 3: 12 months after patients returned their initial FIT (or if they did not return the FIT, 12 months after enrollment) they will be mailed a friendly letter to remind them that it is time for their annual CRC screening and that a FIT kit will be mailed the following week. During the following week the patients will be mailed the FIT kit with addressed stamped envelope and the educational pamphlet they received at enrollment. For follow-up ATR calls, we will use the same protocol as described for the initial screening. Same procedure for year 3.
  automated telephone reminder: The patients will be contacted at 4 weeks and again at 8 weeks if they have not returned the FIT. ATR will remind the patient of the importance of completing and returning the FIT results and encourage screening completion. There will also be an option where the patient can request another FIT kit be mailed to them, one to hear information on common problems with FIT completion or how to call the clinic if they have questions.
- Prevention Coordinator Arm: Years 2 and 3: 12 months after patients returned their initial FIT (or if they did not return the FIT, 12 months after enrollment) they will be mailed a friendly letter to remind them that it is time for their annual CRC screening and that a FIT kit will be mailed the following week. During the following week the patients will be mailed the FIT kit with addressed stamped envelope and the educational pamphlet they received at enrollment. For follow-up PC calls, we will use the same protocol as described for the initial screening. Same procedure for year 3.
  prevention coordinator: The patients will be contacted at 4 weeks and again at 8 weeks if they have not returned the FIT by a prevention coordinator (PC). PC will call to encourage completion and ascertain any barriers to completion. The PCs will use Health Literacy and motivational interviewing techniques described in the training section to enhance understanding and confidence and reduce ambivalence to completing and returning the FIT.
  Annual screening will be further emphasized at enrollment by giving patients an empowering message about the benefits of completing a FIT annually and telling them they will be mailed a reminder letter and FIT kit and receive outreach phone calls in 12 and 24 months for the next two years as well as a post survey and satisfaction interview over the phone at 6 months.
Arm/Group | Automated Telephone Reminder Arm | Prevention Coordinator Arm
Number analyzed (Participants) | 285 | 283
Participants | 104 | 95
Statistical Analysis 1: Comparison: Automated Telephone Reminder Arm vs Prevention Coordinator Arm; Multivariate analyses adjusting for age, race, gender, and health literacy level were done using generalized linear models. A test for interaction between study arm and each of literacy level, age, gender and race was performed to determine whether treatment effect differed by levels of these factors. An unadjusted test for the main effect of each of health literacy level, age, gender, race and study arm was performed to determine whether screening rates differed by levels of these factors; Test type: Superiority; p = 0.30, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Repeat Screening
Description: Patients in our study will be considered to have completed repeat annual CRC screening if they complete a FIT between 12 and 18 months of previous screen (or baseline interview, if initial FIT was not returned). Year 3 primary outcome is number of participants who return a FIT all 3 years.
Time Frame: between 12 and 18 months of previous screen, 2 years overall
Population: 531 eligible for year 3 screening - 614 baseline minus [Year 1 FIT positive (n=44) + Lost to follow-up in year 2 (n=2) + Year 2 FIT positive (n=17) =Lost to follow-up in year 3 (n=20)]
Measure: Count of Participants; unit: Participants
Arm/Group | Automated Telephone Reminder Arm | Prevention Coordinator Arm
Number analyzed (Participants) | 269 | 262
Participants | 58 | 58
Statistical Analysis 1: Comparison: Automated Telephone Reminder Arm vs Prevention Coordinator Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.97, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Prevention Coordinator Arm: Patients will receive Health literacy appropriate education and demonstration of FIT kits with simplified instructions.Patients will receive reminders to complete their FIT screening kits by a prevention coordinator.
  prevention coordinator: The patients will be contacted at 4 weeks and again at 8 weeks if they have not returned the FIT by a prevention coordinator (PC). PC will call to encourage completion and ascertain any barriers to completion. The PCs will use Health Literacy and motivational interviewing techniques described in the training section to enhance understanding and confidence and reduce ambivalence to completing and returning the FIT.
  Years 2 and 3: 12 months after patients returned their initial FIT (or if they did not return the FIT, 12 months after enrollment) they will be mailed a reminder letter and a FIT kit will be mailed the following week. Follow-up procedure will be the same as year 1.
Arm/Group | Automated Telephone Reminder Arm | Prevention Coordinator Arm
All-Cause Mortality (participants affected / at risk) | 0/308 | 1/306
Serious Adverse Events (participants affected / at risk) | 0/308 | 0/306
Other Adverse Events (participants affected / at risk) | 0/308 | 0/306

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT02360605/Prot_SAP_000.pdf